CLINICAL TRIAL: NCT03340142
Title: VIVO™ Accuracy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catheter Precision. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 94-9001-004
Record Dates: First submitted 2017-11-03; First posted 2017-11-13 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Premature Ventricular Contraction; Ventricular Tachycardia
MeSH Terms: conditions — Ventricular Premature Complexes; Tachycardia, Ventricular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): All patients will undergo standard of care ablation procedures. VIVO™ results will be compared to that of standard of care results, but will not be used in diagnosis or treatment.
  Interventions: Device: VIVO™

INTERVENTIONS:
Device: VIVO™ — Diagnose the area of a PVC or VT onset

SUMMARY:
A multi-center study designed to assess the accuracy of VIVO™ in determining the location of a PVC/VT foci in comparison to an electroanatomical mapping system.

DETAILED DESCRIPTION:
The VIVO accuracy study will assess the accuracy of locating a PVC/VT foci by pacing known anatomical locations and comparing the VIVO outcome to that of the Carto system (Biosense-Webster).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are at least 18 years or older
* Subjects who are scheduled for PVC/VT ablation procedure with structurally normal hearts and less than 10% scar.
* Subjects who have signed an IRB/EC approved Informed Consent Form and applicable subject privacy protection authorization per local law
* Subjects will be selected without regard to gender or age (unless precluded by local regulatory requirements)

Exclusion Criteria:

* Subjects who are contraindicated for CT or MRI (must be able to get one)
* Subject whose MRI or CT scan does not comply with the requirements of this protocol
* Subjects who are contraindicated for an electrophysiology procedure and/or fluoroscopy:
* INR > 3
* Active infection
* Pregnancy: Females of childbearing potential with a positive pregnancy test.
* Existing mechanical heart valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-01-29 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of correctly identifying PVC or VT origin | 1 Day
  Determine the accuracy of VIVO in identifying a PVC/VT to the left or right ventricle or the septum. The origin, identified by VIVO, will be compared to the Carto system and the successful ablation location.

SECONDARY OUTCOMES:
Accuracy of correctly identifying known pacing sites | 1 Day
  Determine the accuracy of VIVO in identifying the location of known pacing sites as compared to the Carto system. The origin, identified by VIVO, will be compared to the location identified by Carto as well as the successful ablation location.
Number of adverse events | 1 Day
  Monitor adverse events that occur during the procedure followed by a review from the CEC for correlation to VIVO and adjudication if appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Missiaen Huck, Study Director — Catheter Precision. Inc.
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins Unveristy, Baltimore, Maryland
  - Medical Unversity of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No